CLINICAL TRIAL: NCT05984641
Title: Efficacy and Safety of CONAN® Proctological Cream Formulation in the Topical Treatment of Haemorrhoidal Disease and Anal Fissures: a Randomized Controlled Clinical Trial
Brief Title: Efficacy and Safety of CONAN® Proctological Cream for Treatment of Haemorrhoidal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omikron Italia S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONAN2019
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-08

CONDITIONS: Hemorrhoid Pain; Haemorrhoid Inflammation
Keywords: Haemorrhoids; anal fissures; controlled clinical trial.
MeSH Terms: conditions — Hemorrhoids; Fissure in Ano

STUDY DESIGN:
Intervention Model Description: The study population was randomized into two treatment arms: Group A, active treatment (CONAN® Proctological Cream, Medical Device, Omikron Italia Srl) and Group B, the control group (bowel-function regulation).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Active treatment CONAN® (Medical Device, Omikron Italia Srl) a proctological cream containing 2.5% glycerin macerate from horse chestnut buds (escin), 1% hesperidin, 0.1% hyaluronic acid, 0.1% centella asiatica and 2.5% glycerinic extract of mallow; Instrutction to an healthy diet including an adequate fibre intake and general advice for facilitating evacuation using stool softeners.
  Interventions: Device: CONAN® Proctological Cream
- Group B (No Intervention): No intervention. Instrutction to an healthy diet including an adequate fibre intake and general advice for facilitating evacuation using stool softeners.

INTERVENTIONS:
Device: CONAN® Proctological Cream — The active treatment samples used for the duration of the study were allocated at the site involved and consisted in 30 g tubes with an endorectal applicator, identified by the batch number, expiry date and information on the study on dedicated labels. The treatment of patients randomized to Group A consisted in applying the local treatment (1 application 3 times/day) for 30 days. Instrutction to an healthy diet including an adequate fibre intake and general advice for facilitating evacuation using stool softeners.
  Arms: Group A

SUMMARY:
Aim of the study is to assess the efficacy, safety and tolerability of CONAN® (Proctological Cream, Medical Device, Omikron Italia Srl) on most frequent symptoms in grade 1-2 of haemorrhoidal disease and anal fissures.

DETAILED DESCRIPTION:
Background: To evaluate the role of CONAN® Proctological Cream containing escin, hesperidin and hyaluronic acid in topical treatment of haemorrhoidal disease and anal fissures and its potential efficacy in reducing related symptoms.

Methods: Forty patients with haemorrhoidal disease and anal fissures were enrolled. Of them, 20 were randomized to receive the medical device CONAN® Cream (Group A) and 20 to the untreated control group (Group B). At each scheduled visit, total symptoms were assessed and recorded by assigning a Numerical Rating Scale score from 0 to 10. The adverse events reported by study subjects were also assessed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years
* Hemorrhoidal pathology, anal fissures and anitis
* NRS score ≥ 3 for at least one of the symptoms (burning, itching, feeling of heaviness, foreign body)

Exclusion Criteria:

* Known hypersensitivity to study products
* Proctitis
* Current therapy with other local treatments based on phlebotropes and/or anti-inflammatories
* Surgical treatments undergone less than a year after inclusion
* Pregnancy, breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in the symptom numerical rating scale | 30 days
  The primary outcome was the change in the symptom numerical rating scale (NRS) score after one month (V3) of treatment compared to the baseline in the two groups.

SECONDARY OUTCOMES:
Evaluation of potential adverse events and treatment compliance | 30 days
  The safety of the treatment was investigated by recording and systemic and local adverse events such as systemic allergic reactions, skin sensitisation and discomfort, etc. Treatment compliance was evaluated through assessment by the investigator of the empty study treatment cream tubes returned by patients at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Di Lorenzo, Medicine, Principal Investigator — Department of Surgical Sciences,University of Tor Vergata, Policlinico Tor Vergata; Gabriella Giarratano, Medicine, Study Chair — Department of Surgical Sciences,University of Tor Vergata, Policlinico Tor Vergata
Locations (1):
- Policlinico Tor Vergata Foundation (PTV), Rome, Italy

IPD SHARING:
Plan to Share IPD: No